CLINICAL TRIAL: NCT00478699
Title: Phase III, Open, Multicenter and Randomized Study of Customized Adjuvant Chemotherapy Based on BRCA1 mRNA Levels in Completely Resected Stages II-IIIA Non-Small-Cell Lung Cancer Patients
Brief Title: Randomized Customized Adjuvant Chemotherapy (GECP-SCAT)
Acronym: GECP-SCAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP-SCAT; 2007-000067-15 (EudraCT Number)
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Non-small-cell Lung Cancer
Keywords: SCAT; BRCA1; BRCA1 mRNA Levels; ADJUVANT; LUNG; GECP-SCAT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Control group (Active Comparator): Control group:
  *Docetaxel 75 mg/m2, and cisplatin 75 mg/m2, both on day 1, every 21 days. Total cycles: Four.
  Interventions: Drug: Docetaxel/Cisplatin control
- 2 Experimental group (Experimental): Experimental group, according to the BRAC1 levels of the tumor tissue, will be assigned one of the following treatments:
  * Low expression of BRCA1 → gemcitabine 1250 mg/m2, days 1 and 8, and cisplatin 75 mg/m2, day 1. Cycles every 21 days. Total cycles: 4
  * Intermediate expression levels of BRCA1 → docetaxel 75 mg/m2, and cisplatin 75 mg/m2, both administered on day 1, every 21 days. Total cycles: 4.
  * High expression levels of BRCA1 → docetaxel 75 mg/m2, day 1. Cycles every 21 days. Total cycles: 4.
  Interventions: Drug: Docetaxel; Drug: Gemcitabine/Cisplatin; Drug: Docetaxel/Cisplatin

INTERVENTIONS:
Drug: Docetaxel/Cisplatin control — Docetaxel 75 mg/m2 and cisplatin 75 mg/m2 day 1, 4 cycles
  Other Names: Taxotere/Platinol
  Arms: 1 Control group
Drug: Docetaxel — Docetaxel 75 mg/m2 day 1, 4 cycles
  Other Names: Taxotere
  Arms: 2 Experimental group
Drug: Gemcitabine/Cisplatin — Gemcitabine 1250 mg/m2, day 1 and 8 and cisplatin 75 mg/m2 day 1, 4 cycles
  Other Names: Gemzar/Platinol
  Arms: 2 Experimental group
Drug: Docetaxel/Cisplatin — Docetaxel 75 mg/m2 and cisplatin 75 mg/m2 day 1, 4 cycles
  Other Names: Taxotere/Platinol
  Arms: 2 Experimental group

SUMMARY:
Randomized Study of Customized Adjuvant Chemotherapy based on BRCA1 mRNA Levels in Completely Resected stages II-IIIA Non-Small-Cell Lung Cancer Patients.

DETAILED DESCRIPTION:
Randomized, phase III, predictive pharmacogenomic, open, prospective, international, multicenter study in patients with non-small-cell lung carcinoma (NSCLC) after complete resection and with N1 or N2 involvement

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmation of non-small-cell lung carcinoma.
* Complete surgical resection of the disease.
* Tumoral tissue available for molecular analysis.
* N1 (stage II) or N2 (stage IIIA) lymph node involvement in the study of the operative piece.
* Men or women age 18 years or older.
* Patients with a performance status of 2 or less according to the ECOG classification.
* Patients with the following laboratory results: ANC < 1500/L, Hb < 10 g/dL, platelets <100,000/L, bilirubin < 1.0 mg/dL, AST and ALT < 1.5 upper limit of normality, creatinine clearance < 60 mL/min.
* Complete recovery from surgery within 6 weeks.
* Patients who have given written informed consent before initiating any specific study screening procedure.

Exclusion Criteria:

* Patients who have received previously chemotherapy or radiotherapy for the study disease.
* Impossibility of complying with chemotherapy treatment due to cultural or geographic circumstances.
* Patients with active infection, heart disease, or any other serious disease, in the judgment of the investigator.
* Women who are pregnant or in the period of lactation.
* Patients with a previous diagnosis of malignant disease in the last five years except for carcinoma in situ of the uterine cervix or skin cancer other than melanoma.
* Patients under treatment with investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2007-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bartomeu Massutí Sureda, MD, Study Chair — Hospital General Universitario de Alicante; Jose Miguel Sanchez Torres, MD, Study Chair — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (47):
- Spain (47):
  - Hospital de Elche, Elche, Alicante
  - Ico - H. Germans Trias I Pujol, Badalona, Barcelona
  - Hospital D'Althaia, Manresa, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria, GRAN Canaria
  - Hospital Clin. Univ. Santiago de Compostela, Santiago de Compostela, LA Coruna
  - Hospital San Pedro, Logroño, La Rioja
  - F.H.Alcorcon, Alcorcón, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de La Ribera, Alzira, Valencia
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital de Basurto, Bilbao, Vizcaya
  - H.G.U. Alicante, Alicante
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Univ. Sagrat Cor, Barcelona
  - Instituto Universitario Dexeus, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Ico-Girona (Hospital Josep Trueta), Girona
  - Hospital Virgen de Las Nieves, Granada
  - Hospital de Jaén, Jaén
  - Hospital de León, León
  - Hospital Arnau de Vilanova, Lleida
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital de La Princesa, Madrid
  - Md Anderson Internacional, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital La Paz, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Morales Messeguer, Murcia
  - Clínica Rotger, Palma de Mallorca
  - Hospital Son Dureta, Palma de Mallorca
  - Hospital Son Llátzer, Palma de Mallorca
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital de Donostia, San Sebastián
  - Instituto Oncológico de San Sebastián, San Sebastián
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - H. Arnau de Vilanova, Valencia
  - Hospital General de Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Provincial de Zamora, Zamora
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Lung Cancer Group website — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was 500 patients (intention to treat patient) in 47 centers between June 2007 and May 2013.
Pre-assignment Details: Screening details:
  Experimental arm: according to the BRAC1 levels of the tumor tissue, receive different combination of treatment.
Groups:
- Control Arm: Docetaxel/Cisplatin: Docetaxel 75 mg/m2, and cisplatin 75 mg/m2, both on day 1, every 21 days. Total cycles: 4.
- Experimental Arm: Experimental group, according to the BRAC1 levels of the tumor tissue, one of the following treatments will be assigned:
  * Low expression of BRCA1 gemcitabine 1250 mg / m2, days 1 and 8, and cisplatin 75 mg / m2, day 1. Cycles every 21 days. Total cycles: 4
  * Intermediate expression levels of BRCA1 docetaxel 75 mg / m2, and cisplatin 75 mg / m2, both administered on day 1, every 21 days. Total cycles: 4.
  * High expression levels of BRCA1 docetaxel 75 mg / m2, day 1. Cycles every 21 days. Total cycles: 4.
Period: Overall Study
Arm/Group | Control Arm | Experimental Arm
Started | 108 | 392
Completed | 101 | 355
Not Completed | 7 | 37
Not completed — Inclusion Error | 1 | 7
Not completed — Not receive study treatment | 6 | 30

BASELINE CHARACTERISTICS:
Population: This analisys only include those patients validated by protocol. Patients not valid by protocol will be all those who, having given their informed consent do not receive the study treatment because of any reason and/or those patients who after treatment with chemotherapy do not have a minimum of six months of follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Experimental Arm | Total
Number analyzed (Participants) | 101 | 355 | 456
Age, Continuous [Median (Full Range); unit: years] | 63 [57 to 68] | 61 [56 to 68] | 62 [56 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 74 | 96
  Male | 79 | 281 | 360
Region of Enrollment [Number; unit: participants]
  Spain | 101 | 355 | 456
Smoking habit [Number; unit: participants]
  Former smoker | 62 | 221 | 283
  Smoker | 28 | 102 | 130
  Never smoker | 11 | 32 | 43
Histology [Number; unit: participants]
  Adenocarcinomas | 47 | 175 | 222
  Squamous | 46 | 155 | 201
  Other | 8 | 25 | 33
Staging T [Number; unit: participants] — T: Tumour's Classification by Size
  T1= Tumour < 3 cm in greatest dimension, surrounded by lung or visceral pleura, without bronchoscopic evidence of invasion more proximal than the lobar bronchus T2= Tumour > 3 cm but < 7 cm or tumour
  T3= Tumour > 7 cm or one that directly invades any of the following:
  Chest wall, diaphragm, phrenic nerve, mediastinal pleura, parietal pericardium Tumour in the main bronchus < 2 cm distal to the carina but without involvement of the carina. Associated atelectasis or obstructive pneumonitis of the entire lung Separate tumour nodule(s) in the same lobe
  participants
    T1 | 22 | 68 | 90
    T2 | 64 | 230 | 294
    T3 | 15 | 57 | 72
Staging N [Number; unit: participants] — N: Nodes NX:Regional lymph nodes cannot be assessed N0:No regional lymph node metastasis N1:Metastasis in ipsilateral peribronchial and/or ipsilateral hilar lymph nodes and intrapulmonary nodes, including involvement by direct extension N2:Metastasis in ipsilateral mediastinal and/or subcarinal lymph node(s) N3:Metastasis in contralateral mediastinal, contralateral hilar, ipsilateral or contralateral
  participants
    N1 | 62 | 215 | 277
    N2 | 39 | 140 | 179
Stage [Number; unit: participants] — Staging is a classification where cancer is located, if or where it has spread and whether it's affecting other parts of the body. There are 5 stages for NSCLC (0,I-IV)
  Stage IIA: tumor larger than 4 cm but 5 cm or less in size that hasn't spread to the nearby lymph nodes.
  Stage IIB: tumor that is 5 cm or less in size that has spread to the lymph nodes within the lung, called the N1 lymph nodes. A stage IIB cancer can also be a tumor more than 5 cm wide that has not spread to the lymph nodes.
  Stage III: cancer spread to the lymph nodes but haven't spread to other distant parts of the body
  participants
    IIA | 14 | 38 | 52
    IIB | 37 | 142 | 179
    IIIA | 50 | 175 | 225
Treatment according to BRCA1 level [Number; unit: participants]
  Control: Docetaxel and Cisplatin | 101 | 0 | 101
  Experimental: BRCA1 Low: Gemcitabine / Cisplatin | 0 | 155 | 155
  Experimental BRCA1 medium: Docetaxel / Cisplatin | 0 | 99 | 99
  Experimental BRCA1 High: Docetaxel | 0 | 101 | 101
Treatment compliance [Number; unit: participants]
  Completed | 84 | 307 | 391
  Not completed | 17 | 48 | 65

OUTCOME MEASURES:

1. Primary Outcome: Estimated Overall Survival
Description: To assess and compare the overall survival estimated at 5 years of both treatment groups (Control arm vs Experimental arm).
  Overall survival:The proportion of participants in treatment group who are still alive for a certain period of time after inclusion.
Time Frame: 5 years
Population: Only those patients validated by protocol. Patients not valid by protocol will be all those who, having given their informed consent do not receive the study treatment because of any reason and/or those patients who after treatment with chemotherapy do not have a minimum of six months of follow-up.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 101 | 355
proportion of participants
  Control arm vs Experimental arm | 0.54 [0.44 to 0.64] | 0.56 [0.51 to 0.61]
  Control arm vs Gemcitabine /Cisplatin Experimental arm: number analyzed (Participants) | 101 | 155
  Control arm vs Gemcitabine /Cisplatin Experimental arm | 0.54 [0.44 to 0.64] | 0.56 [0.47 to 0.64]
  Control arm vs Docetaxel /Cisplatin Experimental arm: number analyzed (Participants) | 101 | 99
  Control arm vs Docetaxel /Cisplatin Experimental arm | 0.54 [0.44 to 0.64] | 0.53 [0.42 to 0.62]
  Control arm vs Docetaxel Experimental Arm: number analyzed (Participants) | 101 | 101
  Control arm vs Docetaxel Experimental Arm | 0.54 [0.44 to 0.64] | 0.60 [0.49 to 0.69]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Based on the relevant clinical evidence of the prognostic and predictive value of BRCA1, proposes the present study with which it is intended to demonstrate that adjuvant chemotherapy Individualized based on BRCA1 expression (Experimental arm), it is more effective than chemotherapy without individualize based (Control arm) in patients with completely resected stage II-IIIA NSCLC; Test type: Superiority; p = 0.73, Log Rank; Hazard Ratio (HR) = 0.946, 95% CI 2-sided [0.689 to 1.298]

2. Secondary Outcome: Disease Free Survival
Description: To assess the disease-free survival of both treatment groups. Disease-free survival: will be calculated from the date of surgery until there is some clinical evidence of disease progression or the date of death due to the disease.
Time Frame: 5 years
Population: Participants are analyzed by protocol.
Measure: Median (80% Confidence Interval); unit: Month
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 101 | 355
Month | 38.7 [18.6 to 58.8] | 32.7 [24.1 to 41.2]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Control Arm v Experimental Arm; Test type: Superiority; p = 0.753, Log Rank; Median Difference (Final Values) = 79.3, 95% CI 2-sided [63.5 to 95.1]
Statistical Analysis 2: Comparison: Control Arm vs Experimental Arm; Control Arm v Experimental Arm; Test type: Superiority — The initial hyphotesis were the disease free survival were longest under 65 vs upper 65; p = 0.025, Log Rank; Median Difference (Final Values) = 38.7, 95% CI 2-sided [28 to 38.7]

ADVERSE EVENTS:
Time Frame: 70 month
Groups:
- Control Group: Control group
  - Docetaxel 75 mg/m2, y cisplatin 75 mg/m2, both day 1 every 21 days. Total cycles: 4.
- Experimental Group:All Reported Adverse Events Related to Study Medication: Include participants in experimental arm
  Experimental group, according to the BRAC1 levels of the tumor tissue, will be assigned one of the following treatments:
  * Low expression of BRCA1 → gemcitabine 1250 mg/m2, days 1 and 8, and cisplatin 75 mg/m2, day 1. Cycles every 21 days. Total cycles: 4
  * Intermediate expression levels of BRCA1 → docetaxel 75 mg/m2, and cisplatin 75 mg/m2, both administered on day 1, every 21 days. Total cycles: 4.
  * High expression levels of BRCA1 → docetaxel 75 mg/m2, day 1. Cycles every 21 days. Total cycles: 4.
Arm/Group | Control Group | Experimental Group:All Reported Adverse Events Related to Study Medication
All-Cause Mortality (participants affected / at risk) | 3/108 | 8/392
Serious Adverse Events (participants affected / at risk) | 36/108 | 66/392
Other Adverse Events (participants affected / at risk) | 105/108 | 384/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=108) | Experimental Group:All Reported Adverse Events Related to Study Medication (N=392)
Pulmonary thromboembolism (Vascular disorders) | 2 (2) | 6 (6)
Thrombolysis (Vascular disorders) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 22 (22) | 29 (29)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 14 (14)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anorexy (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Vomits (Gastrointestinal disorders) | 0 (0) | 3 (3)
Acute kidney failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Palmoplantar disease (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 3 (3)
Broken arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than .4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=108) | Experimental Group:All Reported Adverse Events Related to Study Medication (N=392)
Phlebitis (Vascular disorders) | 2 (2) | 9 (9)
Allergic reaction (Immune system disorders) | 1 (1) | 15 (15)
Asthenia (General disorders) | 32 (32) | 266 (266)
Fever (General disorders) | 20 (20) | 20 (20)
Abdominal pain (General disorders) | 6 (6) | 11 (11)
Cardiac disorders (Cardiac disorders) | 2 (2) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 81 (81) | 220 (220)
Leukocites (Blood and lymphatic system disorders) | 8 (8) | 80 (80)
Neutrophils (Blood and lymphatic system disorders) | 5 (5) | 138 (138)
Platelets (Blood and lymphatic system disorders) | 5 (5) | 50 (50)
Epistaxis (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Edema (General disorders) | 2 (2) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 82 (82) | 25 (25)
Sensitivity in sensory processing (Nervous system disorders) | 4 (4) | 47 (47)
Conjunctivitis (Eye disorders) | 2 (2) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 4 (4)
Anorexy (Gastrointestinal disorders) | 11 (11) | 63 (63)
Constipation (Gastrointestinal disorders) | 10 (10) | 57 (57)
Diarrhea (Gastrointestinal disorders) | 20 (20) | 110 (110)
Mucositis (Gastrointestinal disorders) | 5 (5) | 93 (93)
Nausea (Gastrointestinal disorders) | 20 (20) | 180 (180)
Vomiting (Gastrointestinal disorders) | 5 (5) | 126 (126)
Epigastralgia (Gastrointestinal disorders) | 9 (9) | 13 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 142 (142)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 25 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 15 (15)
GGT alteration (Metabolism and nutrition disorders) | 90 (90) | 42 (42)
Creatinine alteration (Metabolism and nutrition disorders) | 10 (10) | 33 (33)
GPT/ GOT alterations (Metabolism and nutrition disorders) | 31 (31) | 37 (37)
LDH alteration (Metabolism and nutrition disorders) | 29 (29) | 29 (29)
Infection (Infections and infestations) | 35 (35) | 51 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No